CLINICAL TRIAL: NCT04351503
Title: A Systems Approach to Predict the Outcome of SARS-CoV-2 in the Population of a City
Brief Title: A Systems Approach to Predict the Outcome of SARS-CoV-2 in the Population of a City; COVID-19
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: sciCORE University of Basel (Unknown); Leonhard Med IT ETH Zurich (Unknown); Swiss Institute of Bioinformatics (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-00769; qu20Egli2
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: SARS Coronavirus (SARS-CoV-2) Infection
Keywords: Coronavirus Disease 2019 (COVID19); SARS-CoV-2 re-infection
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Infections; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SARSCoV-infected patients (cases)
  Interventions: Other: Study A; Other: Study B; Other: Study C; Other: Study D
- non-SARS-CoV-2 infected patients (control): non-SARS-CoV-2 infected patients with or without other respiratory viruses (control).
  Interventions: Other: Study A

INTERVENTIONS:
Other: Study A — Study A: collection of data of clinical outcomes and features of SARS-CoV-2 infection. Demographical, clinical, microbiological, laboratory, epidemiological and hospital-associated data will be analyzed. For this study part, only patients with a visit at the University Hospital Basel will be included in order to access patient charts.
Other: Study B — Study B: collection of epidemiological surveillance data to describe the epidemiology of the SARS-CoV-2 outbreak. The epidemic transmission of Influenza viruses in the City of Basel serves as an important reference to identify similarities and differences to the pandemic SARS-CoV-2 situation. In addition data collected during the Influenza projects - in particular data on statistical blocks of the city, e.g. population density, income and living space will be re-used. Already collected and stored samples such as serum and respiratory material (leftover material) will be (re-) used.
  Groups: SARSCoV-infected patients (cases)
Other: Study C — Study C: data collection for viral evolution. Respiratory materials and matching blood and tissue materials will be used to perform whole genome sequencing to study pathogen evolution between hosts as well as in-host evolution. No additional material will be collected.
  Groups: SARSCoV-infected patients (cases)
Other: Study D — Study D: collection of safety and efficacy data of different treatment modalities. Currently the following treatments are considered as part of the treatment:
  1. Lopinavir/Ritonavir
  2. Hydroxychloroquine
  3. Tocilizumab
  4. Eculizumab
  5. Ruxolitinib
  6. Remdesivir
  7. Treatment with convalescent plasma blood count, blood chemistry and pulmonary function test (collected on a routine basis during hospitalization and in the outpatient setting).
  Groups: SARSCoV-infected patients (cases)

SUMMARY:
This study is to gain critical knowledge to understand the factors influencing the outcome of a pandemic virus within the city of Basel.

DETAILED DESCRIPTION:
In order to evaluate the impact of the new SARS-CoV-2 this study analyzes the clinical outcomes of patients with a confirmed SARS-CoV-2 infection using a systems approach. The objective is to integrate various datasets covering clinical and non-clinical variables. Beside host factors such as age, gender, comorbidities and treatments, microbiological factors, such as SARS-CoV-2 viral loads using a (semi)-quantitative nucleic acid test (QNAT), genome sequences, and virus-specific immune responses are included. In addition, epidemiological aspects within the city, such as case numbers in specific areas and resulting saturation of the healthcare system (e.g. patients being hospitalized, and ICU occupancy), will be analyzed. Further epidemiological data will be generated from biological measurements from all available serum and respiratory samples (leftover material) collected from February 2020 to November 2021 over two seasons as it is likely that a second wave will be circulating in the following winter 2020/2021.

In this project, three retrospective studies will be conducted:

Study A: retrospective observational case-control study to predict the clinical outcomes and features of SARS-CoV-2 infection. The clinical outcomes of SARSCoV-2 infected patients (cases) and non-SARS-CoV-2 infected patients with or without other respiratory viruses (control) will be explored.

Study B: retrospective observational epidemiological surveillance study to describe the epidemiology of the SARS-CoV-2 outbreak; description of the epidemiological spread of the new SARS-CoV-2 virus in people living in Basel.

Study C: retrospective observational viral evolution study whereby respiratory materials and matching blood and tissue materials will be used to perform whole genome sequencing to study pathogen evolution between hosts as well as in-host evolution. No additional material will be collected. Virus genomes obtained during the expanding, peak, and contracting phase of the pandemic will be compared to identify predictors of viral evolution, viral loads, majority species, immune escape variants, and the implications for clinical outcome, diagnostic detection, treatment, and vaccine design. Correlating specifically the occurrence and rate and variants of SARS-CoV-2 re-infections in city blocks of high activity and exposure risk will be of interest.

Study D: retrospective observational treatment outcome study whereby clinical outcome, laboratory, radiological, pulmonary function and virological data as well as data on immune responses will be used to study safety and efficacy of different treatment modalities. All data and material will be collected on a routine basis during hospitalization and in the outpatient setting to assess the safety and effect of different treatment modalities on outcome.

ELIGIBILITY:
Inclusion Criteria:

* Study A: All patients being tested for SARS-CoV-2 at the University Hospital Basel (USB) and with residency in Basel (Basel-Stadt, Riehen, and Bettingen) will be included for clinical outcome evaluation. All age groups will be included. In addition, non-clinical data such as epidemiological and hospital associated data of all people living in Basel but not necessarily tested at the University Hospital Basel will be included
* Study B: Epidemiological data and serum and respiratory samples across all Age groups from people with residency in Basel (Basel-Stadt, Riehen, and Bettingen) with and without confirmed SARS-CoV-2 infection will be included
* Study C: SARS-CoV-2 viral genome analysis will be conducted from all patients tested positive for SARS-CoV-2 genome by NAT at the University Hospital Basel and living in Basel (Basel-Stadt, Riehen, and Bettingen). In addition, viral genome analysis will be conducted from all people tested positive for SARS-CoV-2 genome by NAT living in Basel by the mentioned study partners. All Age groups will be included.
* Patients with cleared SARS-CoV-2 infection coming for plasma donation will be included to describe immunological response after successfully cleared infection.

Exclusion Criteria:

* documented refusal of the general consent or an available/known written or oral statement against Research
* People, who are tested at the USB, with residency outside of Basel (Basel-Stadt, Riehen, and Bettingen)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: SARSCoV- 2 infected patients and non-SARS-CoV-2 infected patients with or without other respiratory viruses with residency in Basel (Basel-Stadt, Riehen, and Bettingen)
Sampling Method: Probability Sample
Enrollment: 126586 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Identification of factors associated with (i) infection (binary, yes/no), (ii) hospitalization (binary, yes/no), (iii) requirement for ICU treatment (binary, yes/no) | at baseline
  Identification of factors associated with (i) infection (binary, yes/no), (ii) hospitalization (binary, yes/no), (iii) requirement for ICU treatment (binary, yes/no)
duration of hospitalization (in days) | at baseline
  duration of hospitalization (in days)
duration of Intensive Care Unit (ICU) stay (in days) | at baseline
  duration of ICU stay (in days)
in-hospital mortality (binary, yes/no) | at baseline
  in-hospital mortality (binary, yes/no)
Number of infected cases within the city of Basel | at baseline
  Number of infected cases confirmed either by nucleic acid test (NAT) or by positive serology within the city of Basel expressed as incidence per statistical block
whole genome sequencing to study pathogen evolution (number, type, and complexity of viral genome) | at baseline
  Number, type, and complexity of viral genome variants and quasispecies identified by deep-sequencing during rise, peak, and contraction of the pandemic in patients and geographic areas.
Identification which treatment modality is associated with adverse events (binary, yes/no) | at baseline
  Identification which treatment modality is associated with adverse events (binary, yes/no)
Identification which treatment modality is associated with pulmonary recovery (binary, yes/no) | after 30 and 90 days
  Identification which treatment modality is associated with pulmonary recovery(binary, yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Egli, Prof. Dr. med., Principal Investigator — Division of Clinical Bacteriology & Mycology, University Hospital Basel
Locations (6):
- Switzerland (6):
  - Viollier AG, Allschwil
  - University Hospital Basel, Basel
  - Biozentrum University of Basel, Basel
  - sciCore University of Basel, Basel
  - Department of Biosystems Science and Engineering ETH Zurich, Basel
  - Swiss Institute of Bioinformatics, Geneva

REFERENCES:
- [Result] Sava M, Sommer G, Daikeler T, Woischnig AK, Martinez AE, Leuzinger K, Hirsch HH, Erlanger T, Wiencierz A, Bassetti S, Tamm M, Tschudin-Sutter S, Stoeckle M, Pargger H, Siegemund M, Boss R, Zimmer G, Vu DL, Kaiser L, Dell-Kuster S, Weisser M, Battegay M, Hostettler K, Khanna N. Ninety-day outcome of patients with severe COVID-19 treated with tocilizumab - a single centre cohort study. Swiss Med Wkly. 2021 Aug 10;151:w20550. doi: 10.4414/smw.2021.20550. eCollection 2021 Aug 2. PMID 34375986
- [Result] Seth-Smith H, Vesenbeckh S, Egli A, Ott S. SARS-CoV-2 in an immunocompromised host: convalescent plasma therapy and viral evolution elucidated by whole genome sequencing. BMJ Case Rep. 2023 Dec 9;16(12):e255255. doi: 10.1136/bcr-2023-255255. PMID 38087481
- [Result] Peter JK, Wegner F, Gsponer S, Helfenstein F, Roloff T, Tarnutzer R, Grosheintz K, Back M, Schaubhut C, Wagner S, Seth-Smith HMB, Scotton P, Redondo M, Beckmann C, Stadler T, Salzmann A, Kurth H, Leuzinger K, Bassetti S, Bingisser R, Siegemund M, Weisser M, Battegay M, Sutter ST, Lebrand A, Hirsch HH, Fuchs S, Egli A. SARS-CoV-2 Vaccine Alpha and Delta Variant Breakthrough Infections Are Rare and Mild but Can Happen Relatively Early after Vaccination. Microorganisms. 2022 Apr 21;10(5):857. doi: 10.3390/microorganisms10050857. PMID 35630302
- [Result] Bruningk SC, Klatt J, Stange M, Mari A, Brunner M, Roloff TC, Seth-Smith HMB, Schweitzer M, Leuzinger K, Sogaard KK, Albertos Torres D, Gensch A, Schlotterbeck AK, Nickel CH, Ritz N, Heininger U, Bielicki J, Rentsch K, Fuchs S, Bingisser R, Siegemund M, Pargger H, Ciardo D, Dubuis O, Buser A, Tschudin-Sutter S, Battegay M, Schneider-Sliwa R, Borgwardt KM, Hirsch HH, Egli A. Determinants of SARS-CoV-2 transmission to guide vaccination strategy in an urban area. Virus Evol. 2022 Mar 17;8(1):veac002. doi: 10.1093/ve/veac002. eCollection 2022. PMID 35310621
- [Derived] Stange M, Mari A, Roloff T, Seth-Smith HM, Schweitzer M, Brunner M, Leuzinger K, Sogaard KK, Gensch A, Tschudin-Sutter S, Fuchs S, Bielicki J, Pargger H, Siegemund M, Nickel CH, Bingisser R, Osthoff M, Bassetti S, Schneider-Sliwa R, Battegay M, Hirsch HH, Egli A. SARS-CoV-2 outbreak in a tri-national urban area is dominated by a B.1 lineage variant linked to a mass gathering event. PLoS Pathog. 2021 Mar 19;17(3):e1009374. doi: 10.1371/journal.ppat.1009374. eCollection 2021 Mar. PMID 33740028